CLINICAL TRIAL: NCT05678660
Title: Study of Neurological Aging Among People Living With HIV (SNAP)
Brief Title: Study of Neurological Aging Among People Living With HIV
Acronym: SNAP
Status: Suspended | Type: Observational
Why Stopped: Due to the release of NIH Policy on Foreign Subawards: NOT-OD-25-104, released on May 1, 2025, funding for this work was suspended pending institution of new procedures. We will resume work as soon as this new procedure is announced.
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Gretchen Birbeck, Professor, University of Rochester
Other Study IDs: RSRB_STUDY00007234; R35NS122265 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2023-01-10 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Aging, Premature
Keywords: frailty; cognitive impairment; neuropathy; mental health; antiretroviral toxicity
MeSH Terms: conditions — Aging, Premature; Frailty; Cognitive Dysfunction; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood sample taken for CD4 count, plasma viral load, and HIV genotyping (about 8mls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Long Group: Older adults individuals with longstanding HIV, stable and on antiretroviral therapy for at least 7 years
- Short Group: Older adults living with HIV, on stable antiretroviral treatment for at least 1 but not more than 2 years,

SUMMARY:
A prospective, exposure-control cohort study of older adults living with HIV comparing the neurological status of those who have had HIV infection for a longer period of time (long HIV group) to age, gender, and community-matched comparison group who have had HIV infection for a shorter period of time (short HIV group).

DETAILED DESCRIPTION:
There is a substantial body of evidence that individuals with long-standing HIV infection experience accelerated neurological aging and prospective lifespan studies that incorporate neuropsychological and imaging outcomes are needed. Elevated risks of cerebrovascular disease are evident throughout the life course of persons living with HIV. Stroke risks are clearly increased in the first few months after antiretroviral initiation. Autopsy studies of adults with HIV 24-48 years of age showed all have vascular changes, specifically lymphocytic perivascular infiltration, thickening of arterial and arteriolar walls, widened perivascular space, hypertrophy of the vascular muscle layers and perivascular amyloid deposition. Even when excluding individuals with a history of stroke, cerebrovascular disease risk factors are associated with decreased cognitive capacity in persons with HIV. Basal ganglia enhancement on MRI indicative of decreased regional cerebral blood flow and blood brain barrier breakdown is associated with HIV dementia.

HIV-associated neurocognitive disorder is another manifestation of accelerated aging. Using diffusion tensor imaging and data from healthy controls to calculate an "brain age gaps" in individuals with HIV infection, the "brain age gap", is associated with plasma viral load and cognitive function. In an autopsy study comparing HIV+ persons age 36-60 years with age-matched controls, HIV showed increased amyloid beta immunostaining. The accumulation of these proteins may be one possible mechanisms of accelerated aging in HIV. Some have proposed that BBB breakdown secondary to vascular dysfunction may contribute to this deposition. Distal sensory polyneuropathy (DSPN), a common neurological comorbidity in HIV that also increases in frequency with age in HIV negative individuals. Despite extensive diagnostic evaluations, ~40% of people with a DSPN will have no clear underlying cause identified. DSPN is more common and complex in African population with additional underlying etiologies being medication toxicities and nutritional deficiencies.In the RAAZ study, investigators identified a high prevalence of DSPN among HIV infected individuals prior to ART initiation which is associated with low body mass index and food insecurity. More recent neuropathy studies have shown that folate deficiency may play a role in DSPN in Zambia with HIV+ individuals being especially susceptible. Epilepsy incidence shows a bimodal age distribution with the increased incidence of seizures and epilepsy in the elderly attributed to the increase of age-related and aging-related epileptogenic conditions. While the overall prevalence of epilepsy can be expected to increase with advanced age in HIV, identifying risk factors for this among persons for epilepsy among those with controlled systemic disease may offer important insights into the pathophysiology.

HIV-associated accelerated aging of the nervous system is thought to be related to ongoing low grade inflammation in the setting of treated HIV. Poor CNS penetration of some antiretroviral therapies (ARVs) has also been proposed as one problem contributing to neurological morbidity in systemically controlled HIV. ARV neurotoxicity is also important. Multiple studies have highlighted both the short and long term neurotoxicity of efavirenz. Darunavir and ritonavir may increase the risk of aging-related cerebral degeneration. Heneka 2020 proposed that COVID survivors may be at increased risk of neurological disorders due to direct negative effects of SARS-CoV-2, acceleration of pre-existing problems or de novo induction of neurodegenerative process. Poor complex motor performance in persons with HIV is associated with higher inflammatory burden. A recent report from Ghana found stroke admissions and mortality rates have increased since SARS-CoV-2's arrival.

In the SNAP Study, the investigators will utilize the existing consortia of neuro-HIV rural study sites to enroll 150 HIV+ adults >45 years of age stable on ARVs for at least 7 years and an age, gender, and community-matched comparison group of HIV+ adults stable on ARVs for 1-2 years. These individuals will undergo annual assessments for 6 years to evaluate their general and neurological health and the aging process that evolves during the 6 years of assessments.

Understanding whether or not PLWH experience accelerated aging of the nervous system will provide critical insights for health services planning as antiretroviral therapies allow PLWH to live into middle and late years. Identifying risk factors for specific neurologic aging issues will guide clinical care and screening and may inform regarding the pathophysiological mechanisms involved including the possibility that some therapies contribute to the long-term neurotoxicity of the condition.

ELIGIBILITY:
Inclusion Criteria:

* For the short group, stable on ART for 1 year, but no more than 2 years.
* For long group, on ART for 7 or more years

Exclusion Criteria:

* Acute medical illness.
* Decisional impairment precluding informed consent as noted by clinicians providing care to the patient or by the research staff team members.
* Communication impairments-unable to hear or unable to speak.
* Being unable to communicate in English or in the dominant language at the study site (Tonga).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified through the antiretroviral clinics associated with Chikankata Hospital and Monze Mission Hospital in Zambia's Southern Province. Individuals will first be identified in the long group and will then be matched to a PLWH in the short group matching based upon gender, age and community of residents
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2028-06-05 (Estimated); Study Completion 2028-06-05 (Estimated)

PRIMARY OUTCOMES:
Cognition - Zambian Mini-Mental Status Examination (zMMSE) - During enrollment | baseline/during enrollment
  The zMMSE is an adaptation of the well-known MMSE which provides single summary score with a maximum of 30 points
Cognition - Zambian Mini-Mental Status Examination (zMMSE) - on Year 1 of evaluation | Year 1 evaluation
  The zMMSE is an adaptation of the well-known MMSE which provides single summary score with a maximum of 30 points
Cognition - Zambian Mini-Mental Status Examination (zMMSE) - on Year 2 of evaluation | Year 2 evaluation
  The zMMSE is an adaptation of the well-known MMSE which provides single summary score with a maximum of 30 points
Cognition - International HIV Dementia Scale (I-HDS) - on Year 3 of evaluation | Year 3 evaluation
  The IHDS assesses registration, recall, motor speed and psychomotor speed and provides a single summary score of a maximum of 12 points
Cognition - International HIV Dementia Scale (I-HDS)- on Year 4 of evaluation | Year 4 evaluations
  The IHDS assesses registration, recall, motor speed and psychomotor speed and provides a single summary score of a maximum of 12 points
Cognition - International HIV Dementia Scale (I-HDS) - on Year 5 of evaluation | Year 5 evaluation
  The IHDS assesses registration, recall, motor speed and psychomotor speed and provides a single summary score of a maximum of 12 points
Cognition - International HIV Dementia Scale (I-HDS)- on Year 6 of evaluation | Year 6 evaluation
  The IHDS assesses registration, recall, motor speed and psychomotor speed and provides a single summary score of a maximum of 12 points
Mental Health - The Alcohol Use Disorders Identification Test (AUDIT) -Baseline/during enrollment | Baseline/during enrollment
  The Alcohol Use Disorders Identification Test (AUDIT) is an alcohol screening instrument for patient self reporting. This 10-item alcohol screen helps identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). A score of 1 to 7 =low-risk consumption; 8 to 14 suggest harmful alcohol consumption, and ≥15 moderate-severe alcohol use disorder with a total score of 40.
Mental Health - The Alcohol Use Disorders Identification Test (AUDIT) - on Year 1 of enrollment | Year 1 evaluation
  The Alcohol Use Disorders Identification Test (AUDIT) is an alcohol screening instrument for patient self reporting. This 10-item alcohol screen helps identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). A score of 1 to 7 =low-risk consumption; 8 to 14 suggest harmful alcohol consumption, and ≥15 moderate-severe alcohol use disorder with a total score of 40.
Mental Health - The Alcohol Use Disorders Identification Test (AUDIT)- on year 2 of evaluation | Year 2 evaluation
  The Alcohol Use Disorders Identification Test (AUDIT) is an alcohol screening instrument for patient self reporting. This 10-item alcohol screen helps identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). A score of 1 to 7 =low-risk consumption; 8 to 14 suggest harmful alcohol consumption, and ≥15 moderate-severe alcohol use disorder with a total score of 40.
Mental Health - The Alcohol Use Disorders Identification Test (AUDIT) - on year 3 of evaluation | Year 3 evaluation
  The Alcohol Use Disorders Identification Test (AUDIT) is an alcohol screening instrument for patient self reporting. This 10-item alcohol screen helps identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). A score of 1 to 7 =low-risk consumption; 8 to 14 suggest harmful alcohol consumption, and ≥15 moderate-severe alcohol use disorder with a total score of 40.
Mental Health - Center for Epidemiologic Studies Depression Scale (CES-D)- on year 4 of evaluation | Year 4 evaluation
  is a 7-item screen with a total score for the seven items ranging from 0 to 21. In most populations, 0-4: minimal anxiety / 5-9: mild anxiety / 10-14: moderate anxiety/ 15-21: severe anxiety.
Mental Health - Center for Epidemiologic Studies Depression Scale (CES-D)- on year 5 of evaluation | Year 5 evaluation
  is a 7-item screen with a total score for the seven items ranging from 0 to 21. In most populations, 0-4: minimal anxiety / 5-9: mild anxiety / 10-14: moderate anxiety/ 15-21: severe anxiety.
Mental Health - Center for Epidemiologic Studies Depression Scale (CES-D)- on year 6 of evaluation | Year 6 evaluation
  is a 7-item screen with a total score for the seven items ranging from 0 to 21. In most populations, 0-4: minimal anxiety / 5-9: mild anxiety / 10-14: moderate anxiety/ 15-21: severe anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- baseline/during enrollment | Baseline
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- baseline/during enrollment | Baseline/during enrollment
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- on year 1 of evaluation | Year 1 evaluation
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- on year 2 of evaluation | Year 2 evaluation
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- on year 3 of evaluation | Year 3 evaluation
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- on year 4 of evaluation | Year 4 evaluation
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- on year 5 of evaluation | Year 5 evaluation
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - The Generalized Anxiety Disorders Screen (GAD-7)- on year 6 of evaluation | Year 6 evaluation
  General Anxiety Disorder-7 (GAD-7). GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. The higher the score, the more severe the anxiety.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ)-baseline/during enrolment | Baseline/during enrollment
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ)- on year 1 of enrolment | Year 1 evaluation
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ)- on year 1 of evaluation | Year 2 evaluation
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ)- on year 3 of evaluation | Year 3 evaluation
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ)- on year 4 of evaluation | Year 4 evaluation
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ)- on year 5 of evaluation | Year 5 evaluation
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Mental Health - An adaptation of the Harvard Trauma Questionnaire (HTQ) - on year 6 of evaluation | Year 6 evaluation
  Includes 10 traumatic events yielding a score of 0-10 and then 40 follow-up questions regarding post traumatic symptoms that will be delivered only to individuals scoring at least 1 on the initial 10 questions. The post traumatic symptom score will range is from 0-120.
Frailty assessment - Body weight - baseline/during enrollment | Baseline/during enrollment
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurement: Body weight in kilograms (kg).
Frailty assessment - Body weight - on year 1 of evaluation. | Year 1 evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurements: Body Weight in kilograms (kg)
Frailty assessment - Body weight- on year 2 of evaluation | Year 2 evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurements: Body Weight in kilograms (kg)
Frailty assessment - Body weight - on year 3 of evaluation | Year 3 evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurements: Body Weight, Body Fat, Body Muscle, and the Body Mass Index (BMI).
Frailty assessment - Body weight on year 4 of evaluation | Year 4 evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurements: Body Weight in kilograms(kg)
Frailty assessment - Body weight - on year 5 | Year 5 evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurements: Body Weight, Body Fat, Body Muscle, and the Body Mass Index (BMI).
Frailty assessment - Body weight - on year 6 of evaluation | Year 6 evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the following measurements: Body Weight in kilograms(kg).
Frailty assessment - Body height- baseline/during enrollment | Baseline/during enrollment
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body height- on year 1 of evaluation | Year 1 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body height- on year 2 of evaluation | Year 2 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body height- on year 3 of evaluation | Year 3 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body height- on year 4 of evaluation | Year 4 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body height- on year 5 of evaluation | Year 5 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body height- on year 6 of evaluation | Year 6 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The height scale will be used to capture height in meters (m).
Frailty assessment - Body mass index-baseline/during enrollment | Baseline/during enrollment
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessment - Body mass index- on year 1 of evaluation | Year 1 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessment - on year 2 of evaluation | Year 2 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessment - Body mass index- on year 3 of evaluation | Year 3 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessment - Body mass index- on year 4 of evaluation | Year 4 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessment - Body mass index- on year 5 of evaluation | Year 5 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessment - Body mass index- on year 6 of evaluation | Year 6 of evaluation
  Body composition describes percentages of fat, bone, and muscle in the human body. Body composition also represents a more accurate description of weight and provides a better understanding of the overall health of an individual. Measuring body composition is part of the frailty assessment. The smart scale will be used to capture a full body composition analysis, which includes the Body Mass Index (BMI) in kilograms(kg). With the following interpretation below 18.5 - underweight range. between 18.5 and 24.9 - healthy weight range. between 25 and 29.9 - overweight range. between 30 and 39.9 - obese range.
Frailty assessments - Grip strength- baseline/during enrollment | Baseline
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frailty assessments - Grip strength - on year 1 of evaluation | Year 1 evaluation
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frailty assessments - Grip strength- on year 2 of evaluation | Year 2 evaluation
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frailty assessments - Grip strength- on year 3 of evaluation | Year 3 evaluation
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frailty assessments - Grip strength- on year 4 of evaluation | Year 4 evaluation
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frailty assessments - Grip strength-on year 5 of evaluation | Year 5 evaluation
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frailty assessments - Grip strength- on year 6 of evaluation | Year 6 evaluation
  Grip strength will be assessed by dynamometry against international norms for age and SNAP_Protocol_V2.3_14June22 Page 7 of 12 Version Date: 2.3 14June22 gender and will be classified as weak, normal or strong.
Frail assessment - Physical Activity- baseline/during enrollment | Baseline
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Physical Activity- on year 1 of evaluation | Year 1 evaluation
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Physical Activity- on year 2 of evaluation | Year 2 evaluation
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Physical Activity- on year 3 of evaluation | Year 3 evaluation
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Physical Activity- on year 4 of evaluation | Year 4 evaluation
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Physical Activity- on year 5 of evaluation | Year 5 evaluation
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Physical Activity- on year 6 of evaluation | Year 6 evaluation
  Physical activity will be scored from 0-100 based upon will be determined based upon self-report in response to a list of items of commonly undertaken activities in this population.
Frail assessment - Time Gait- baseline/during enrollment | baseline
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Frail assessment - Time Gait- on year 1 of evaluation | Year 1 evaluation
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Frail assessment - Time Gait- on year 2 of evaluation | Year 2 evaluation
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Frail assessment - Time Gaiton year 3 of evaluation | Year 3 evaluation
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Frail assessment - Time Gait- on year 4 of evaluation | Year 4 evaluation
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Frail assessment - Time Gait- on year 5 of evaluation | Year 5 evaluation
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Frail assessment - Time Gait- on year 6 of evaluation | Year 6 evaluation
  Gait speed is based upon a 15-foot times gait. Normative walking speeds are not available in this population, but decline over time (in the same participant) and comparison within the matched pair will be used to determine slowed gait.
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- baseline/during enrollment | baseline/ during enrollment
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- on year 1 of evaluation | Year 1 of evaluation
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- on year 2 of evaluation | Year 2 evaluation
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- on year 3 of evaluation | Year 3 evaluation
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- on year 4 of evaluation | Year 4 evaluation
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- on year 5 of evaluation | Year 5 evaluation
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Brief Peripheral Neuropathy (BPNS)- on year 6 of evaluation | Year 6 evaluation
  The brief peripheral neuropathy screen yields a dichotomous outcome (neuropathy present vs absent).
Peripheral nerve health - Heart Rate Variability(HRV)- baseline/during enrollment | Baseline/during enrollment
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.
Peripheral nerve health - Heart Rate Variability(HRV)- on year 1 of evaluation | Year 1 evaluation
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.
Peripheral nerve health - Heart Rate Variability(HRV) - on year 2 of evaluation | Year 2 evaluation
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.
Peripheral nerve health - Heart Rate Variability(HRV)- on year 3 of evaluation | Year 3 evaluation
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.
Peripheral nerve health - Heart Rate Variability(HRV)- on year 4 of enrollment | Year 4 evaluation
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.
Peripheral nerve health - Heart Rate Variability(HRV)- on year 5 of evaluation | Year 5 evaluation
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.
Peripheral nerve health - Heart Rate Variability(HRV)- on year 6 of evaluation | Year 6 evaluation
  Heart rate variability will measure autonomic function. Baseline heart rate will be assessed and a heart rate variability score produced with higher scores generally representing better autonomic function. Comparisons between the two groups and the individual participants HRV trajectory over time will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L. Birbeck, MD, Principal Investigator — University of Rochester
Locations (3):
- Zambia (3):
  - Chilenje Level 1 Hospital, Lusaka, Lusaka Province
  - Chikankata Hospital, Mazabuka, Southern Province
  - Monze Mission Hospital, Monze, Southern Province

IPD SHARING:
Plan to Share IPD: Yes
Access to databases and associated software tools generated under the project will be available for educations, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 2 years after study completion
Access Criteria: Written request

REFERENCES:
- [Background] Mbewe EG, Kabundula PP, Mwanza-Kabaghe S, Buda A, Adams HR, Schneider C, Potchen MJ, Mweemba M, Mathews M, Menon JA, Wang B, Baseler T, Paciorkowski A, Birbeck GL, Bearden DR. Socioeconomic Status and Cognitive Function in Children With HIV: Evidence From the HIV-Associated Neurocognitive Disorders in Zambia (HANDZ) Study. J Acquir Immune Defic Syndr. 2022 Jan 1;89(1):56-63. doi: 10.1097/QAI.0000000000002825. PMID 34878435
- [Background] Bearden DR, Omech B, Rulaganyang I, Sesay SO, Kolson DL, Kasner SE, Mullen MT. Stroke and HIV in Botswana: A prospective study of risk factors and outcomes. J Neurol Sci. 2020 Jun 15;413:116806. doi: 10.1016/j.jns.2020.116806. Epub 2020 Mar 26. PMID 32244092
- [Background] Dean O, Buda A, Adams HR, Mwanza-Kabaghe S, Potchen MJ, Mbewe EG, Kabundula PP, Moghaddam SM, Birbeck GL, Bearden DR. Brain Magnetic Resonance Imaging Findings Associated With Cognitive Impairment in Children and Adolescents With Human Immunodeficiency Virus in Zambia. Pediatr Neurol. 2020 Jan;102:28-35. doi: 10.1016/j.pediatrneurol.2019.08.014. Epub 2019 Sep 9. PMID 31604645
- [Background] Heneka MT, Golenbock D, Latz E, Morgan D, Brown R. Immediate and long-term consequences of COVID-19 infections for the development of neurological disease. Alzheimers Res Ther. 2020 Jun 4;12(1):69. doi: 10.1186/s13195-020-00640-3. PMID 32498691
- [Background] Kvalsund M, Kayamba V, Kelly P, Birbeck GL, Mwansa-Thurman C, Sommer IN, Lamers Y, Gardiner J, Herrmann DN. Is folate deficiency a common cause of distal symmetric polyneuropathy in Zambian clinics? J Neurol Sci. 2020 Feb 15;409:116583. doi: 10.1016/j.jns.2019.116583. Epub 2019 Nov 20. PMID 31864072
- [Background] Monreal E, Gullon P, Perez-Torre P, Escobar-Villalba A, Acebron F, Quereda Rodriguez-Navarro C, Sanchez-Ruano L, Fernandez-Felix BM, Muriel A, Perez-Elias MJ, Masjuan J, Corral I. Increased HIV infection in patients with stroke in Spain. A 16-year population-based study. Enferm Infecc Microbiol Clin (Engl Ed). 2020 May;38(5):219-225. doi: 10.1016/j.eimc.2019.10.006. Epub 2019 Dec 16. English, Spanish. PMID 31859019
- [Background] Sarfo FS, Mensah NO, Opoku FA, Adusei-Mensah N, Ampofo M, Ovbiagele B. COVID-19 and stroke: Experience in a Ghanaian healthcare system. J Neurol Sci. 2020 Sep 15;416:117044. doi: 10.1016/j.jns.2020.117044. Epub 2020 Jul 16. PMID 32702560
- [Background] Barrell K, Smith AG. Peripheral Neuropathy. Med Clin North Am. 2019 Mar;103(2):383-397. doi: 10.1016/j.mcna.2018.10.006. Epub 2018 Dec 17. PMID 30704689
- [Background] Feinstein MJ, Hsue PY, Benjamin LA, Bloomfield GS, Currier JS, Freiberg MS, Grinspoon SK, Levin J, Longenecker CT, Post WS. Characteristics, Prevention, and Management of Cardiovascular Disease in People Living With HIV: A Scientific Statement From the American Heart Association. Circulation. 2019 Jul 9;140(2):e98-e124. doi: 10.1161/CIR.0000000000000695. Epub 2019 Jun 3. PMID 31154814
- [Background] Hammond CK, Eley B, Ing N, Wilmshurst JM. Neuropsychiatric and Neurocognitive Manifestations in HIV-Infected Children Treated With Efavirenz in South Africa-A Retrospective Case Series. Front Neurol. 2019 Jul 9;10:742. doi: 10.3389/fneur.2019.00742. eCollection 2019. PMID 31338063
- [Background] Kuhn T, Jin Y, Huang C, Kim Y, Nir TM, Gullett JM, Jones JD, Sayegh P, Chung C, Dang BH, Singer EJ, Shattuck DW, Jahanshad N, Bookheimer SY, Hinkin CH, Zhu H, Thompson PM, Thames AD. The joint effect of aging and HIV infection on microstructure of white matter bundles. Hum Brain Mapp. 2019 Oct 15;40(15):4370-4380. doi: 10.1002/hbm.24708. Epub 2019 Jul 4. PMID 31271489
- [Background] Lin HL, Muo CH, Lin CY, Chen HJ, Chen PC. Incidence of stroke in patients with HIV infection: A population-based study in Taiwan. PLoS One. 2019 May 22;14(5):e0217147. doi: 10.1371/journal.pone.0217147. eCollection 2019. PMID 31116762
- [Background] Mapoure Njankouo Y, Mondomobe Atchom C, Halle MP, Mbatchou Ngahane BH, Luma NH. Prevalence of HIV infection among stroke patients in Douala. Med Sante Trop. 2019 May 1;29(2):184-189. doi: 10.1684/mst.2019.0895. PMID 31379346
- [Background] Montoya JL, Campbell LM, Paolillo EW, Ellis RJ, Letendre SL, Jeste DV, Moore DJ. Inflammation Relates to Poorer Complex Motor Performance Among Adults Living With HIV on Suppressive Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2019 Jan 1;80(1):15-23. doi: 10.1097/QAI.0000000000001881. PMID 30365450
- [Background] Pluta A, Wolak T, Sobanska M, Gawron N, Egbert AR, Szymanska B, Horban A, Firlag-Burkacka E, Bienkowski P, Sienkiewicz-Jarosz H, Scinska-Bienkowska A, Desowska A, Rusiniak M, Biswal BB, Rao S, Bornstein R, Skarzynski H, Lojek E. HIV and age underlie specific patterns of brain abnormalities and cognitive changes in high functioning patients. Neuropsychology. 2019 Mar;33(3):358-369. doi: 10.1037/neu0000504. Epub 2019 Jan 28. PMID 30688492
- [Background] Beghi E, Giussani G. Aging and the Epidemiology of Epilepsy. Neuroepidemiology. 2018;51(3-4):216-223. doi: 10.1159/000493484. Epub 2018 Sep 25. PMID 30253417
- [Background] Benjamin L, Khoo S. HIV infection and stroke. Handb Clin Neurol. 2018;152:187-200. doi: 10.1016/B978-0-444-63849-6.00015-3. PMID 29604976
- [Background] Cross HM, Chetty S, Asukile MT, Hussey HS, Lee Pan EB, Tucker LM. A proposed management algorithm for late-onset efavirenz neurotoxicity. S Afr Med J. 2018 Mar 28;108(4):271-274. doi: 10.7196/SAMJ.2017.v108i4.12914. PMID 29629676
- [Background] Gordon SB, Chinula L, Chilima B, Mwapasa V, Dadabhai S, Mlombe Y; Malawi Research Ethics Workshop 2018 Participants. A Malawi guideline for research study participant remuneration. Wellcome Open Res. 2018 Dec 19;3:141. doi: 10.12688/wellcomeopenres.14668.2. eCollection 2018. PMID 30662959
- [Background] Kvalsund M, Chidumayo T, Hamel J, Herrmann D, Heimburger D, Peltier A, Birbeck G. Factors associated with distal symmetric polyneuropathies in adult Zambians: A cross-sectional, observational study of the role of HIV, non-antiretroviral medication exposures, and nutrition. J Neurol Sci. 2018 May 15;388:61-69. doi: 10.1016/j.jns.2018.02.035. Epub 2018 Feb 22. PMID 29627032
- [Background] Seden K, Kiiza D, Laker E, Arinaitwe WJ, Waitt C, Lamorde M, Khoo S. High prevalence and long duration of nervous system and psychiatric adverse drug reactions in Ugandan patients taking efavirenz 600 mg daily. J Antimicrob Chemother. 2018 Nov 1;73(11):3158-3161. doi: 10.1093/jac/dky298. PMID 30085168
- [Background] Soontornniyomkij V, Umlauf A, Soontornniyomkij B, Gouaux B, Ellis RJ, Levine AJ, Moore DJ, Letendre SL. Association of antiretroviral therapy with brain aging changes among HIV-infected adults. AIDS. 2018 Sep 10;32(14):2005-2015. doi: 10.1097/QAD.0000000000001927. PMID 29912063
- [Background] Dickens AM, Yoo SW, Chin AC, Xu J, Johnson TP, Trout AL, Hauser KF, Haughey NJ. Chronic low-level expression of HIV-1 Tat promotes a neurodegenerative phenotype with aging. Sci Rep. 2017 Aug 10;7(1):7748. doi: 10.1038/s41598-017-07570-5. PMID 28798382
- [Background] Kuhn T, Schonfeld D, Sayegh P, Arentoft A, Jones JD, Hinkin CH, Bookheimer SY, Thames AD. The effects of HIV and aging on subcortical shape alterations: A 3D morphometric study. Hum Brain Mapp. 2017 Feb;38(2):1025-1037. doi: 10.1002/hbm.23436. Epub 2016 Oct 25. PMID 27778407
- [Background] Nookala AR, Mitra J, Chaudhari NS, Hegde ML, Kumar A. An Overview of Human Immunodeficiency Virus Type 1-Associated Common Neurological Complications: Does Aging Pose a Challenge? J Alzheimers Dis. 2017;60(s1):S169-S193. doi: 10.3233/JAD-170473. PMID 28800335
- [Background] Sandkovsky U, Podany AT, Fletcher CV, Owen A, Felton-Coleman A, Winchester LC, Robertson K, Swindells S. Impact of efavirenz pharmacokinetics and pharmacogenomics on neuropsychological performance in older HIV-infected patients. J Antimicrob Chemother. 2017 Jan;72(1):200-204. doi: 10.1093/jac/dkw403. Epub 2016 Sep 21. PMID 27655857
- [Background] Cysique LA, Brew BJ. The effects of HIV and aging on brain functions: proposing a research framework and update on last 3 years' findings. Curr Opin HIV AIDS. 2014 Jul;9(4):355-64. doi: 10.1097/COH.0000000000000078. PMID 24871088
- [Background] Andras IE, Toborek M. Amyloid beta accumulation in HIV-1-infected brain: The role of the blood brain barrier. IUBMB Life. 2013 Jan;65(1):43-9. doi: 10.1002/iub.1106. Epub 2012 Dec 7. PMID 23225609
- [Background] Cettomai D, Kwasa JK, Birbeck GL, Price RW, Cohen CR, Bukusi EA, Kendi C, Meyer AC. Screening for HIV-associated peripheral neuropathy in resource-limited settings. Muscle Nerve. 2013 Oct;48(4):516-24. doi: 10.1002/mus.23795. Epub 2013 Aug 27. PMID 24037693
- [Background] Chang L, Holt JL, Yakupov R, Jiang CS, Ernst T. Lower cognitive reserve in the aging human immunodeficiency virus-infected brain. Neurobiol Aging. 2013 Apr;34(4):1240-53. doi: 10.1016/j.neurobiolaging.2012.10.012. Epub 2012 Nov 15. PMID 23158761
- [Background] Benjamin LA, Bryer A, Emsley HC, Khoo S, Solomon T, Connor MD. HIV infection and stroke: current perspectives and future directions. Lancet Neurol. 2012 Oct;11(10):878-90. doi: 10.1016/S1474-4422(12)70205-3. PMID 22995692
- [Background] Birbeck GL, Kvalsund MP, Byers PA, Bradbury R, Mang'ombe C, Organek N, Kaile T, Sinyama AM, Sinyangwe SS, Malama K, Malama C. Neuropsychiatric and socioeconomic status impact antiretroviral adherence and mortality in rural Zambia. Am J Trop Med Hyg. 2011 Oct;85(4):782-9. doi: 10.4269/ajtmh.2011.11-0187. PMID 21976587
- [Background] Harezlak J, Buchthal S, Taylor M, Schifitto G, Zhong J, Daar E, Alger J, Singer E, Campbell T, Yiannoutsos C, Cohen R, Navia B; HIV Neuroimaging Consortium. Persistence of HIV-associated cognitive impairment, inflammation, and neuronal injury in era of highly active antiretroviral treatment. AIDS. 2011 Mar 13;25(5):625-33. doi: 10.1097/QAD.0b013e3283427da7. PMID 21297425
- [Background] Clark US, Cohen RA. Brain dysfunction in the era of combination antiretroviral therapy: implications for the treatment of the aging population of HIV-infected individuals. Curr Opin Investig Drugs. 2010 Aug;11(8):884-900. PMID 20721831
- [Background] Foley J, Ettenhofer M, Wright MJ, Siddiqi I, Choi M, Thames AD, Mason K, Castellon S, Hinkin CH. Neurocognitive functioning in HIV-1 infection: effects of cerebrovascular risk factors and age. Clin Neuropsychol. 2010 Feb;24(2):265-85. doi: 10.1080/13854040903482830. PMID 20162495
- [Background] Kandiah PA, Atadzhanov M, Kvalsund MP, Birbeck GL. Evaluating the diagnostic capacity of a single-question neuropathy screen (SQNS) in HIV positive Zambian adults. J Neurol Neurosurg Psychiatry. 2010 Dec;81(12):1380-1. doi: 10.1136/jnnp.2009.183210. Epub 2010 Jun 11. PMID 20543182
- [Background] Achim CL, Adame A, Dumaop W, Everall IP, Masliah E; Neurobehavioral Research Center. Increased accumulation of intraneuronal amyloid beta in HIV-infected patients. J Neuroimmune Pharmacol. 2009 Jun;4(2):190-9. doi: 10.1007/s11481-009-9152-8. Epub 2009 Mar 17. PMID 19288297
- [Background] Birbeck GL, Chomba E, Kvalsund M, Bradbury R, Mang'ombe C, Malama K, Kaile T, Byers PA, Organek N; RAAZ Study Team. Antiretroviral adherence in rural Zambia: the first year of treatment availability. Am J Trop Med Hyg. 2009 Apr;80(4):669-74. PMID 19346397
- [Background] Chang L, Wong V, Nakama H, Watters M, Ramones D, Miller EN, Cloak C, Ernst T. Greater than age-related changes in brain diffusion of HIV patients after 1 year. J Neuroimmune Pharmacol. 2008 Dec;3(4):265-74. doi: 10.1007/s11481-008-9120-8. Epub 2008 Aug 15. PMID 18709469
- [Background] Chomba E, Haworth A, Atadzhanov M, Mbewe E, Birbeck GL. The socioeconomic status of children with epilepsy in Zambia: implications for long-term health and well-being. Epilepsy Behav. 2008 Nov;13(4):620-3. doi: 10.1016/j.yebeh.2008.06.008. Epub 2008 Aug 12. PMID 18602496
- [Background] Sacktor NC, Wong M, Nakasujja N, Skolasky RL, Selnes OA, Musisi S, Robertson K, McArthur JC, Ronald A, Katabira E. The International HIV Dementia Scale: a new rapid screening test for HIV dementia. AIDS. 2005 Sep 2;19(13):1367-74. PMID 16103767
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Goodkin K, Wilkie FL, Concha M, Hinkin CH, Symes S, Baldewicz TT, Asthana D, Fujimura RK, Lee D, van Zuilen MH, Khamis I, Shapshak P, Eisdorfer C. Aging and neuro-AIDS conditions and the changing spectrum of HIV-1-associated morbidity and mortality. J Clin Epidemiol. 2001 Dec;54 Suppl 1:S35-43. doi: 10.1016/s0895-4356(01)00445-0. PMID 11750208
- [Background] 44. WHO. The Alcohol Use Disorders Identification Test 2nd edition. Online: WHO; 2001: http://www.who.int/substance_abuse/publications/en/.
- [Background] Berger JR, Nath A, Greenberg RN, Andersen AH, Greene RA, Bognar A, Avison MJ. Cerebrovascular changes in the basal ganglia with HIV dementia. Neurology. 2000 Feb 22;54(4):921-6. doi: 10.1212/wnl.54.4.921. PMID 10690987
- [Background] Dufouil C, Clayton D, Brayne C, Chi LY, Dening TR, Paykel ES, O'Connor DW, Ahmed A, McGee MA, Huppert FA. Population norms for the MMSE in the very old: estimates based on longitudinal data. Mini-Mental State Examination. Neurology. 2000 Dec 12;55(11):1609-13. doi: 10.1212/wnl.55.11.1609. PMID 11113212
- [Background] Fazeka F, Ropele S, Bammer R, Kapeller P, Stollberger R, Schmidt R. Novel imaging technologies in the assessment of cerebral ageing and vascular dementia. J Neural Transm Suppl. 2000;59:45-52. doi: 10.1007/978-3-7091-6781-6_7. PMID 10961417
- [Background] Izycka-Swieszewska E, Zoltowska A, Rzepko R, Gross M, Borowska-Lehman J. Vasculopathy and amyloid beta reactivity in brains of patients with acquired immune deficiency (AIDS). Folia Neuropathol. 2000;38(4):175-82. PMID 11693722
- [Background] Roberts RE, Vernon SW. The Center for Epidemiologic Studies Depression Scale: its use in a community sample. Am J Psychiatry. 1983 Jan;140(1):41-6. doi: 10.1176/ajp.140.1.41. PMID 6847983